CLINICAL TRIAL: NCT01041898
Title: The Bone-Fat-Pancreas Axis in Children: Establishing a Role for Undercarboxylated Osteocalcin in Energy Homeostasis
Brief Title: The Bone-Fat-Pancreas Axis in Children
Status: Completed | Type: Observational
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Krista Casazza, Assistant Professor, University of Alabama at Birmingham
Other Study IDs: F091118001
Record Dates: First submitted 2009-12-30; First posted 2010-01-01 (Estimated); Last update posted 2019-11-25 (Actual); Status verified 2019-11

CONDITIONS: Bone Mineral Density; Body Fat Distribution; Insulin Homeostasis
Keywords: osteocalcin; insulin; body composition; bone mineral density; Evaluate the effect of osteocalcin on bone mineral density; Evaluate the effect of osteocalcin on body fat distribution; Evaluate the effect of osteocalcin on insulin homeostasis
MeSH Terms: conditions — Insulin Resistance

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Samples will be labeled with the study protocol number, a unique identifier, and the date of collection.
  Specimens will be obtained by the nursing staff at the PCIR. The PCIR processing lab will process the samples, which will then be stored in a locked freezer at -80oC in the restricted access CNRU Metabolism Core lab (WEBB 337).
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The overarching hypothesis of this proposal is that obesity and positive energy balance in children promote both low bone mass accrual and risk for diabetes through events that are mechanistically associated and that involve bone as an endocrine organ. Recent studies conducted in mice have uncovered the presence of a unique "bone-fat-pancreas" axis that regulates energy homeostasis, coordinates energy partitioning between bone and adipose tissue, and impacts insulin sensitivity. The adipocyte-derived hormone leptin, elevated levels of which reflect both adiposity and positive energy balance, inhibits bone formation via sympathetic activation. Decreased bone formation in turn depresses insulin sensitivity and secretion via decreased production of undercarboxylated osteocalcin (unOC), a novel bone-derived hormone. Although data from mice are compelling, this novel pathway has not been widely tested in humans. Sparse data from adult men and women suggest that this axis is active in humans, and that unOC is regulated in part by exercise. No data are available regarding the bone-fat-pancreas axis in children. Because the foundations of body composition trajectories and metabolic "programming" are established early in the life course, childhood, particularly during early stages of growth and development, is an especially salient time period for evaluating the bone-fat-pancreas axis. With this pilot grant, we propose to gather evidence that these interrelationships exist in children. The data from this project will be used to prepare an NIH R01 proposal to conduct a lifestyle-based intervention in children aimed both at reducing risk for osteoporosis and type 2 diabetes, and at identifying the role of unOC in metabolism and tissue partitioning.

Hypothesis 1: Obesity and positive energy balance in children decrease bone mass via elevated leptin.

Specific Aim 1: Determine the association between bone mass by DXA and serum leptin concentration in lean and obese children. We predict that body weight will be positively associated with bone mass, but that at any given body weight, bone mass will be lower in obese children, and that this difference will be explained by leptin.

Hypothesis 2: Leptin-mediated suppression of unOC decreases insulin secretion through action on the β-cell, and decreases insulin sensitivity by inhibiting secretion of adiponectin from adipose tissue.

Specific Aim 2: Determine the association between insulin secretion during oral glucose tolerance test (OGTT; from C-peptide modeling) and serum unOC in lean and obese children. Determine the association between insulin sensitivity during OGTT (derived from mathematical modeling) and serum unOC in lean and obese children. Obese children are less insulin sensitive, and in an absolute sense, secrete more insulin. However, we predict that at any given degree of insulin sensitivity, insulin secretion will be lower in obese children, and that this difference will be explained by unOC. unOC will be inversely associated with serum leptin, and will be positively associated with adiponectin and insulin sensitivity.

Hypothesis 3: Physical activity prevents leptin suppression of unOC and partitions energy towards bone mineral at the expense of bone marrow adipose tissue.

Specific Aim 3: Assess the interrelationships among physical activity using accelerometry, bone mass using DXA and bone marrow adipose tissue using magnetic resonance imaging. We predict that at any given level of serum leptin, active children will have greater unOC. Further, we predict that at any given body weight, active children will have greater bone mass and lesser bone marrow adipose tissue than inactive children.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Self-identified as European American (Caucasian) of African American
* Aged 5 to 10 years
* Healthy, not under the care of a doctor
* Not taking medications known to affect body composition or metabolism
* Pre-pubertal

Exclusion Criteria:

* Not meeting above criteria

Ages: 5 Years to 10 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Healthy European American (Caucasian) girls aged five to ten years
Sampling Method: Non-Probability Sample
Enrollment: 28 (Actual)
Dates: Start 2009-12; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Evaluate the role of undercarboxylated osteocalcin on body composition and insulin homeostasis | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Krista Casazza, PhD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- UAB, Birmingham, Alabama, United States